CLINICAL TRIAL: NCT06133751
Title: Effect of 8-week Supplementation With Anthocyanin Compounds Contained in Black Chokeberry on Inflammation and Oxidative Stress Induced by Very Intense Exercise in Highly Trained Rowers
Brief Title: Effect of 8-week Supplementation With Black Chokeberry on Recovery in Highly Trained Rowers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Poznan University of Physical Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: SKaczmarczyk_PhD
Record Dates: First submitted 2023-10-27; First posted 2023-11-15 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2023-10

CONDITIONS: Inflammation;Muscle(S); Oxidative Stress Injury; Permeability; Increased
MeSH Terms: conditions — Myositis, Inclusion Body

STUDY DESIGN:
Intervention Model Description: Participants randomly divided into one of two groups. The supplemented group (n=7) receives chokeberry capsules, while the control group (n=8) receives a placebo product.
Who Masked: Participant
Masking Description: Youth National Rowing Team of Poland
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplemented group (Experimental): Athletes in the supplemented group (n=7) consumed capsules with highly concentrated 18% chokeberry extract. One capsule contained 200 mg. In addition to chokeberry extract, each capsule also contained chokeberry fiber, E460b magnesium salts of stearic acid (anti-caking agent), E551 silicon dioxide (anti-caking agent), hydroxypropyl methylcellulose (capsule shell) and E171 titanium dioxide (shell color).
  The rowers (both supplemented and control group) took 3 capsules a day (at breakfast, lunch and dinner) for 8 weeks. The athletes sipped each capsule with a glass of water.
  Interventions: Drug: black chokeberry (Aronia melanocarpa)
- Placebo group (Placebo Comparator): The control group (n=8) consumed capsules that were made from chokeberry fiber.
  The rowers (both supplemented and control group) took 3 capsules a day (at breakfast, lunch and dinner) for 8 weeks. The athletes sipped each capsule with a glass of water.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: black chokeberry (Aronia melanocarpa) — Black chokeberry capsules standardized for anthocyanin compounds
  Arms: Supplemented group
Drug: Placebo — Chokeberry fiber placebo capsules
  Arms: Placebo group

SUMMARY:
Purpose: To analyze the effects of 8-week supplementation with anthocyanin compounds contained in black chokeberry (Aronia melanocarpa) on indicators of inflammation and oxidative stress.

Hypothesis: Supplementation with anti-inflammatory and antioxidant anthocyanin compounds improves recovery from intense exercise by reducing inflammation and oxidative stress in highly trained rowers

The study consisted of a nutritional intervention (supplementation) - with compounds of natural origin - chokeberry extract (capsules) - 18% standardized for anthocyanin content (dose 3 x 200 mg per day) - that is, 107 mg of pure anthocyanins per day, or a placebo product that was made from chokeberry fiber

Study plan I term of the study

1. Conduct a body composition analysis, body height, food diary, self reported gastrointestinal scale
2. Collection of blood samples before the exercise test for biochemical determinations.
3. Exercise test of 2000m on a rowing ergometer.
4. Collection of blood immediately after exercise and 1 hours after
5. Collection of blood for biochemical determinations 24 hours after the end of the exercise test
6. Supplementation for 8 weeks 2nd test date Repeat the measurements from the 1st test date.

Participants: Youth National Rowing Team of Poland Experimental procedure: Observation of the effect of black chokeberry consumption on parameters of inflammation, oxidative stress and intestinal parameters during the immediate start preparation period in highly skilled rowers.

DETAILED DESCRIPTION:
Participants Twenty participants from the Youth National Rowing Team of Poland have been recruited for the study. In the end, fifteen rowers participated in the study (two did not show up for the first date, three more were absent for the second date). Before the first and second dates of the study, a body composition analysis was performed using the TANITA MC-780 with an accuracy of 0.05 kg, and hight was measured throughout sea 217 hightmeter. The experiment was conducted in accordance with the Declaration of Helsinki. The study protocol was approved by the Ethical Committee of the Medical University of Poznan (resolution no. 390/22). All players were informed of the exact course of the study and gave written consent to participate.

Youth National Rowing Team of Poland The athletes' diets were completely analyzed before each exercise test by a nutritionist. Participants, with the help of a dietician who was available during meals on test days, filled out food diaries. The amount of energy, protein, carbohydrates, fats and fiber were then analyzed using a commercially available program.

Experimental procedure The rowers were randomly divided into two groups-supplemented and control, it was a double-blind study. Athletes in the supplemented group (n=7) consumed capsules with highly concentrated 18% chokeberry extract. One capsule contained 200 mg. In addition to chokeberry extract, each capsule also contained chokeberry fiber, E460b magnesium salts of stearic acid (anti-caking agent), E551 silicon dioxide (anti-caking agent), hydroxypropyl methylcellulose (capsule shell) and E171 titanium dioxide (shell color). The control group (n=8) consumed capsules that were made from chokeberry fiber. All additional substances the same as in capsules with chokeberry extract. The supplement and placebo product was manufactured by MBL BIOTRADE, Poznań. The rowers (both supplemented and control group) took 3 capsules a day (at breakfast, lunch and dinner) for 8 weeks. The athletes sipped each capsule with a glass of water.

Exercise test On two testing dates (before and after supplementation), the athletes performed a 2,000-meter test on a rowing ergometer (Concept II, USA). Athletes had to complete the test in the shortest possible time overcoming the maximum load. The results of the test were taken into account in the selection for the championship team so the athletes performed the task with great motivation. Before the test, each competitor individually performed a 5-minute warm-up.

Material collection and examination Samples were taken at three time points: pre (before the exercise test) post (immediately after the exercise test and 1 hour after) and recovery (24 hours after the exercise test) both before and after the supplementation period. Blood samples were collected from the elbow vein into 9-ml tubes (to obtain serum) and centrifuged at 3,000 rpm and into 2.7-ml tubes (to determine morphology). Morphology was determined on the same day the samples were collected, while serum was frozen and stored at -80oC until assays were performed. In addition, before and immediately after the exercise test, capillary blood was drawn from the earlobe to determine lactate levels.

Measurements TAC (Total Antioxidant Capacity), TBARS (levels of lipid peroxidation products), IL-2, IL-6, IL-10, TNF-α and myoglobin levels were determined using ELISA kits (SunRed Biotechnology Company). Lactate levels were determined immediately after capillary blood sampling using a commercially available kit (Dr. Lange, Germany). The concentration of lactate was determined in mmol/l. intestinal parameters: LBP (lipopolysacharide-binding pro), Claudin3, I-FABP (intestinal fatty acid binding pro). After both tests, participants filled out self-reported gastrointestinal scale.

Any data obtained during the research will be used only for the purposes of this research project. The participant has the right to access and correct his/her data, to obtain information regarding the processing of his/her personal data, to request the deletion or restriction of the processing of his/her data, the right to portability of the data provided, the right to object to the processing, and the right to withdraw consent to the processing of personal data at any time. Withdrawal of consent does not affect the lawfulness of processing carried out on the basis of consent before its withdrawal.

The confidential nature of the research documentation will be respected throughout the study. Legal requirements for the protection of personal data will be observed. In the study documentation, participants will be identified by a nadem code at the beginning of the study. The results of this study will be published after pooled data analysis. Thus, the identity of the participants will remain confidential.

The place of data storage is the university's branch office in Gorzow Wielkopolski.

All parameters will be analyzed using Elisamtests and read on the ELISAMAR reader. In terms of statistical measures, the following will be performed: descriptive statistics, Shapiro-Wilk test to assess normality, and multivariate analysis of variance ANOVA test.

ELIGIBILITY:
Inclusion Criteria:

* Training experience a minimum of five years
* Minimum training time per week 240 minute
* Membership in the Youth National Rowing Team of Poland
* Completion of the 2000m ergometer test on two test dates

Exclusion Criteria:

* Taking other supplements containing anthocyanin compounds during the study period or a month earlier
* Antibiotic therapy
* Health problems

Ages: 18 Years to 24 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-06-10 (Actual); Study Completion 2023-06-10 (Actual)

PRIMARY OUTCOMES:
Level of total antioxidants (TAC) | 8 weeks
  ELISA kits (SunRed Biotechnology Company) - Indicators of pro-oxidant-antioxidant balance
interleukins: IL-2, IL-6, IL-10 | 8 weeks
  ELISA kits (SunRed Biotechnology Company) - Immunological indicators
lactic acid | 8 weeks
  Diaglobal, Berlin, Germany)
LBP (lipopolysacharide-binding pro) | 8 weeks
  ELISA kits (SunRed Biotechnology Company) - Gut parameter
level of lipid peroxidation products (TBARS) | 8 weeks
  ELISA kits (SunRed Biotechnology Company) - Indicators of pro-oxidant-antioxidant balance
(NO) nitric oxide | 8 weeks
  obtained by indirect method Griessa - Indicators of pro-oxidant-antioxidant balance
comet assay (DNA damage) | 8 weeks
  comet assay BioTechne
tumor necrosis factor (TNF α) | 8 weeks
  ELISA kits (SunRed Biotechnology Company) - Immunological indicators
myoglobin | 8 weeks
  ELISA kits (SunRed Biotechnology Company)
I-FABP (intestinal fatty acid binding protein) | 8 weeks
  ELISA kits (SunRed Biotechnology Company) - Gut parameter
Claudin3 | 8 weeks
  ELISA kits (SunRed Biotechnology Company) - Gut parameter

SECONDARY OUTCOMES:
gastrointestinal symptom scale | 8 weeks
  Self-reported 10-point scale, 10 is the most severe symptoms on the scale
energy [kcal] | 8 weeks
  dietitian program
protein [g] | 8 weeks
  dietitian program
fat [g] | 8 weeks
  dietitian program
carbohydrate [g] | 8 weeks
  dietitian program
fiber [g] | 8 weeks
  dietitian program
body hight [m] | 8 weeks
  secco 217 highmeter
body mass [kg] | 8 weeks
  body analyzer
body fat [%,kg] | 8 weeks
  body analyzer
total body water [%,kg] | 8 weeks
  body analyzer
lean body mass [kg] | 8 weeks
  body analyzer

CONTACTS AND LOCATIONS:
Overall Officials: Anna Skarpańska-Stejnborn, Professor, Study Director — Poznan University of Physical Education
Locations (1):
- University of Physical Education in Poznan, Poznan, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kaczmarczyk S, Kasperska A, Dziewiecka H, Ostapiuk-Karolczuk J, Cichon-Wozniak J, Basta P, Skarpanska-Stejnborn A. A single 2000-meter exercise test to assess exercise adaptation in elite rowers during the preparatory phase. Front Physiol. 2025 Aug 12;16:1544637. doi: 10.3389/fphys.2025.1544637. eCollection 2025. PMID 40873756